CLINICAL TRIAL: NCT02416765
Title: An Open-label, Randomized, Five-way, Cross-over Study to Compare the Efficacy of Single- and Dual-hormone Closed-loop Operations Combined With Either Conventional Carbohydrate Counting or a Simplified Qualitative Meal-size Estimation, and Sensor-augmented Pump Therapy in Regulating Glucose Levels in Adults With Type 1 Diabetes
Brief Title: Closed-loop Control of Postprandial Glucose Levels in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, MD, PhD, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS10
Record Dates: First submitted 2015-04-02; First posted 2015-04-15 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop strategy; Artificial pancreas; Postprandial glucose; Insulin; Glucagon; Hypoglycemia; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Hypoglycemia | interventions — Methods; Insulin; Insulin Lispro; Insulin Aspart; Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sensor-augmented pump therapy (Active Comparator): Patients will use conventional pump therapy and freely implement their usual basal rate and CHO-matching full prandial bolus to regulate glucose levels.
  Interventions: Other: 15-hour intervention
- Single-hormone CLS with full boluses (Active Comparator): Variable subcutaneous insulin infusion rates will be used to regulate postprandial glucose levels. Carbohydrate-matching full prandial bolus will be given 10 minutes before the meal. Each subject insulin-to-carbohydrate ratio will be used to calculate the insulin bolus to be given.
  Interventions: Other: 15-hour intervention; Drug: Insulin (Lispro, Aspart or guilisine); Other: Closed-loop strategy
- Single-hormone CLS with partial boluses (Active Comparator): Variable subcutaneous insulin infusion rates will be used to regulate postprandial glucose levels. A pre-meal partial prandial bolus will be given 10 minutes before the meal. The partial bolus will be based on the estimated meal size (snack-regular-large-very large). Meal size will be defined as: snack as any meal less than 30g, regular meal as any meal between 30g and 60g CHO, large meal as any meal between 60g and 90g CHO, very large meal for anything above 90g CHO.
  Interventions: Other: 15-hour intervention; Drug: Insulin (Lispro, Aspart or guilisine); Other: Closed-loop strategy
- Dual-hormone CLS with full boluses (Active Comparator): Variable subcutaneous insulin and glucagon infusion rates will be used to regulate postprandial glucose levels. Carbohydrate-matching full prandial bolus will be given 10 minutes before the meal. Each subject insulin-to-carbohydrate ratio will be used to calculate the insulin bolus to be given.
  Interventions: Other: 15-hour intervention; Drug: Insulin (Lispro, Aspart or guilisine); Drug: Glucagon (Eli Lilly); Other: Closed-loop strategy
- Dual-hormone CLS with partial boluses (Active Comparator): Variable subcutaneous insulin and glucagon infusion rates will be used to regulate postprandial glucose levels. A pre-meal partial prandial bolus will be given 10 minutes before the meal. The partial bolus will be based on the estimated meal size (snack-regular-large-very large). Meal size will be defined as: snack as any meal less than 30g, regular meal as any meal between 30g and 60g CHO, large meal as any meal between 60g and 90g CHO, very large meal for anything above 90g CHO.
  Interventions: Other: 15-hour intervention; Drug: Insulin (Lispro, Aspart or guilisine); Drug: Glucagon (Eli Lilly); Other: Closed-loop strategy

INTERVENTIONS:
Other: 15-hour intervention — Interventions will be conducted in outpatient settings. Subject's usual insulin will be used. Meals will not be standardized. Subjects will be allowed to eat whatever and when they want and will be allowed to drink alcohol. Subjects will be allowed to exercise, but they will be asked to do the same amount and intensity of exercise on all intervention visits. Subjects will be accompanied all the time by a member from the research team during closed-loop visits to implement hormonal infusions.
Drug: Insulin (Lispro, Aspart or guilisine) — Patient's usual insulin (Lispro, Aspart or guilisine) will be used in all interventions.
  Arms: Dual-hormone CLS with full boluses; Dual-hormone CLS with partial boluses; Single-hormone CLS with full boluses; Single-hormone CLS with partial boluses
Drug: Glucagon (Eli Lilly) — In the dual-hormone CLS interventions, glucagon (Eli Lilly) will be used.
  Arms: Dual-hormone CLS with full boluses; Dual-hormone CLS with partial boluses
Other: Closed-loop strategy — Every 10 minutes, the glucose level as measured by the real time sensor (Dexcom G4 Platinum, Dexcom) will be entered manually into the computer. The pumps' infusion rate will then be changed manually based on the computer generated recommendation infusion rates. The computer generated recommendations are based on a predictive algorithm.
  Arms: Dual-hormone CLS with full boluses; Dual-hormone CLS with partial boluses; Single-hormone CLS with full boluses; Single-hormone CLS with partial boluses

SUMMARY:
Postprandial meal glucose control with closed-loop systems (CLS) still needs some improvements. In the postprandial period, sensor delay in detecting blood glucose rise after a meal together with delays in insulin absorption expose patients to early risk of hyperglycemia and then to late-postprandial hypoglycemia. Glucagon infusion in dual-hormone CLS has the potential to improve post-meal control as compared to single-hormone CLS allowing a better glucose excursion related to a more aggressive insulin infusion while minimizing hypoglycemic risk. Several approaches have been tested for the determination of prandial boluses during closed-loop operation.

The objective of this study is to test in outpatient unrestricted settings whether, in the context of closed-loop strategy, conventional meal carbohydrate counting could be reduced to a simplified qualitative meal size estimation without a significant degradation in overall glycemic control in adult patients with type 1 diabetes.

The investigators hypothesize that in outpatient free-living conditions: 1) Dual-hormone CLS with partial boluses is equivalent to dual-hormone CLS with full boluses in terms of mean glucose; 2) Single-hormone CLS with partial boluses is equivalent to single-hormone CLS with full boluses in terms of mean glucose. Secondary hypothesis are: 3) Dual-hormone CLS with partial boluses will decrease time in hypoglycemia compared to single-hormone CLS with partial boluses; 4) Dual-hormone CLS with partial boluses is better than sensor-augmented pump therapy in terms of mean glucose; 5) Single-hormone CLS with partial boluses is better than sensor-augmented pump therapy in terms of mean glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months and currently using a fast actin insulin analog (Lispro, Aspart or Guilisine).
4. Last (less than 3 months) HbA1c ≤ 10%.
5. Currently using carbohydrate counting as the meal insulin dose strategy.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Ongoing pregnancy.
4. Severe hypoglycemic episode within 1 month of screening.
5. Agents affecting gastric emptying (Motilium®, Prandase®, Victoza®, Byetta® and Symlin®) as well as oral anti-diabetic agents (Metformin, SGLT-2 inhibitors and DPP-4 inhibitors) if not at a stable dose for 3 months. Otherwise, these medications are acceptable and will be kept stable during the entire protocol.
6. Oral steroids unless patients present a low stable dose (e.g. 10 mg or less of prednisone per day or physiological doses, less than 35 mg/day, of hydrocortisone Cortef®). Inhale steroids at stable dose in the last month are acceptable.
7. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator (e.g. unstable psychiatric condition).
8. Failure to comply with team's recommendations (e.g. not willing to change pump parameters, follow algorithm's suggestions, etc).
9. Living or planned travel outside Montreal (> 1h of driving) area during closed-loop procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mean glucose levels as measured by the glucose sensor. | 15 hours
  The following comparisons will be done: 1) Dual-hormone CLS with partial boluses vs. dual-hormone CLS with full boluses; 2) Single-hormone CLS with partial boluses vs. single-hormone CLS with full boluses.

SECONDARY OUTCOMES:
Mean glucose levels as measured by the glucose sensor | 15 hours
  The following comparisons will be done: 1) Dual-hormone CLS with partial boluses vs. single-hormone CLS with partial boluses; 2) Dual-hormone CLS with partial boluses vs. sensor-augmented pump therapy; 3) Single-hormone CLS with partial boluses vs. sensor-augmented pump therapy.
Percentage of time of sensor glucose concentrations between 4 and 8 mmol/L | 15 hours
Percentage of time of sensor glucose concentrations between 4 and 10 mmol/L | 15 hours
Percentage of time of sensor glucose concentrations above 10 mmol/L | 15 hours
Percentage of time of sensor glucose concentrations above 14 mmol/L | 15 hours
Percentage of time of glucose levels spent below 4 mmol/L | 15 hours
Percentage of time of glucose levels spent below 3.1 mmol/L | 15 hours
Area under the curve of glucose values below 4 mmol/L | 15 hours
Area under the curve of glucose values below 3.1 mmol/L | 15 hours
Number of patients with at least one hypoglycemic event below 3.1 mmol/L with or without symptoms | 15 hours
Total number of hypoglycemic event below 3.1 mmol/L | 15 hours
Total insulin delivery | 15 hours
Total glucagon delivery | 15 hours
Standard deviation of glucose levels | 15 hours
Total carbohydrate intake | 15 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada